CLINICAL TRIAL: NCT03367533
Title: Alpha-Amino-3-Hydroxy-5-Methyl-4- Isoxazole Propionic Acid Receptor Components of the Anti-Depressant Ketamine Response
Brief Title: Alpha-Amino-3-Hydroxy-5-Methyl-4- Isoxazole Propionic Acid Receptor Components of the Anti-Depressant Ketamine Response, Pilot Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2000021345; No NIH funding per PI (Other: CB 9.20.23)
Record Dates: First submitted 2017-11-14; First posted 2017-12-08 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Depressive Disorder, Major; Post Traumatic Stress Disorder; Bipolar Disorder
Keywords: Depression; Ketamine; Magnetic Resonance Imaging
MeSH Terms: conditions — Depressive Disorder, Major; Stress Disorders, Post-Traumatic; Bipolar Disorder; Depression | interventions — Ketamine; perampanel

STUDY DESIGN:
Intervention Model Description: The investigators employ a counter-balanced cross-over design in which ketamine plus perampanel is given on one day, and approximately 21 days later ketamine plus placebo is given.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ketamine plus perampanel (Experimental): A screening session is conducted to ensure that the subject can safely receive perampanel and ketamine (physical exam, blood and urine analyses, electrocardiogram, drug and alcohol testing). The participant will then receive 6 milligrams (mg) oral perampanel and intravenous ketamine. Participants will then undergo a 2-hour magnetic resonance imagining (MRI) scan. The following day, participants will return for an additional scan and symptom assessment.
  Interventions: Drug: Ketamine; Drug: Perampanel
- ketamine plus placebo (Placebo Comparator): A screening session is conducted to ensure that the subject can safely receive perampanel and ketamine (physical exam, blood and urine analyses, electrocardiogram, drug and alcohol testing). The participant will then receive an oral placebo (in lieu of 6 mg oral perampanel) and intravenous ketamine. Participants will then undergo a 2-hour MRI scan. The following day, participants will return for an additional scan and symptom assessment.
  Interventions: Drug: Ketamine; Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — Intravenous ketamine
Drug: Perampanel — Oral perampanel (6 mg)
  Arms: ketamine plus perampanel
Drug: Placebo — Oral placebo
  Arms: ketamine plus placebo

SUMMARY:
The proposed study will assess the combined effect of perampanel and ketamine on the anti-depressant response in individuals with treatment resistant depression. The purpose of this study is to test the hypothesis that stimulation of Alpha-Amino-3-Hydroxy-5-Methyl-4- Isoxazole Propionic Acid receptors (AMPAR) is critical to the anti-depressant response of ketamine.

DETAILED DESCRIPTION:
The proposed study is the first in humans to assess the necessity of Alpha-Amino-3-Hydroxy-5-Methyl-4- Isoxazole Propionic Acid receptors (AMPAR) stimulation for the emergence of the anti-depressant effects of ketamine. Despite the overall safety and efficacy of ketamine, concerns remain. For example, ketamine is a drug with abuse liability. Similarly, it produces transient cognitive and perceptual changes that are distressing for some patients. Therefore, it is critical to determine which aspects of ketamine's effects on neural systems. To do this, we employ perampanel, an FDA-approved drug that blocks calcium and non-calcium dependent AMPARs. We employ a counter-balanced cross-over design in which ketamine plus perampanel is given on one day, and approximately 21 days later ketamine plus placebo is given. The effects of these drug combinations are assessed via fMRI studies of neural functional connectivity and oxidative metabolism as well as interview and self-report measures on the infusion day and 24 hours later. If perampanel blocks the capacity of ketamine to ameliorate the clinical and neural signatures of major depression, it would suggest that AMPAR stimulation is critical for the anti- depressant effects of ketamine in humans. This would support the further exploration of drugs that selectively enhance the stimulation of AMPARs without blocking N-methyl-D-aspartate receptors (NMDARs), such as AMPAkines and metabotropic glutamate receptor 2 (mGluR2) antagonists as anti-depressants.

Specific hypotheses include:

The purpose of this study is to test the hypothesis that stimulation of Alpha-Amino-3-Hydroxy-5-Methyl-4- Isoxazole Propionic Acid receptors (AMPAR) is critical to the anti-depressant response of ketamine.

Specifically, we will test the following hypotheses:

1. Perampanel pre-treatment reduces ketamine-related increases in prefrontal functional connectivity and CMRO2 during ketamine infusion in individuals with treatment-resistant depression.
2. Perampanel pre-treatment reduces ketamine-induced increases in prefrontal CMRO2 and functional connectivity observed at 24 hours in individuals with treatment resistant depression.
3. Perampanel pre-treatment reduces the positive effect of ketamine on clinical improvement as measured by the Hamilton Depression Inventory (1) at 24 hours in individuals with treatment resistant depression.

Exploratory: Changes in prefrontal functional connectivity and CMRO2 during ketamine infusion and 24 hours post-infusion are correlated with clinical improvement as measured by the Hamilton Depression Inventory in individuals with treatment resistant depression.

As this study is the first, to the investigator's knowledge, to involve using ketamine and perampanel in human subjects, the investigators have included a small out-of-scanner study to test the safety of the ketamine/perampanel combination on 3 healthy subjects. This registration focuses on the main study that will follow the safety evaluation and evaluate the effect of perampanel and ketamine on individuals with treatment resistant depression.

ELIGIBILITY:
Inclusion Criteria Substudy #2:

* Participants between the ages of 18-65
* Right-handed as determined by the Edinburgh Handedness Inventory
* Current depression as indicated by a score greater than 17 on the full Hamilton Depression Rating Scale
* Anti-depressant resistant depressive symptoms, defined by a history of failure of one or more adequate anti-depressant trials
* Individuals who have previously received ketamine must have had a positive response. Individuals who report reduced depressive symptoms will be treated as ketamine responders and entered directly into the closed label trial.
* Participants will meet DSM-5 Criteria for MDD, Bipolar or PTSD as determined by the SCID-5
* All participants given ketamine must be engaged in treatment outside of the research protocol. Those who are not currently in treatment may be referred for treatment.
* Individuals who are receiving pharmacotherapy for depression must have been receiving the current medication and dose for 4 weeks before randomization. In addition, they should have a plan to continue the current regime of pharmacotherapy for the duration of the trial.
* Individuals who are receiving psychotherapy must have been in treatment for four weeks and should have a plan to continue the current regime of psychotherapy for the duration of the trial.
* Willing to refrain from caffeine, drug and alcohol use for one week prior to each MRI session
* Females will be included if they are not pregnant or breastfeeding and agree to utilize a medically accepted birth control method (to include oral, injectable, or implant birth control, condom, diaphragm with spermicide, intrauterine device, tubal ligation, abstinence, or partner with vasectomy). Women who are surgically sterile or post-menopausal with cessation of menses for at least one year are not required to use birth control. If a woman should become pregnant during the study, she will be excluded from the trial.
* Females will receive ketamine during the follicular phase, i.e., in the first week after the start of the menstrual period, if at all possible. If a prospective participant typically has significant menstrual cramps during this entire follicular phase, she will be studied during another part of her cycle. She will be studied during the same part of her cycle for each scan, if possible.
* Able to read and write English
* Have at least a 12th grade education level or equivalent

Exclusion Criteria Substudy #2:

* A score on the Columbia Suicide Severity Rating Scale in the "intent" or "intent with plan" categories or judged by Dr. Krystal or Dr. Driesen to be at serious risk for suicide.
* Neurological disorder excluding migraine headaches or more than mild head injury. Individuals with migraines will not complete any ketamine infusion visits within 24 hours of a migraine. More than mild head injury is indicated by the presence of any of the following:

  * More than half hour unconsciousness after trauma
  * More than one hour post-traumatic amnesia
  * Concussive symptoms such as headache, memory problems, nausea/vomiting, irritability, ringing in the ears, dizziness, balance problems, difficulty concentrating or visual disturbances lasting more than one week after injury.
  * Concussive symptoms as defined above in the first week after injury causing more than one day impairment in typical duties.
  * Four or more concussive events of less severity than the above will also be grounds for exclusion. These events would include post-trauma symptoms such as the individual being dazed, seeing stars, unconscious for less than one half hour, or post-traumatic amnesia of less than an hour.
* Current therapeutic treatment with ketamine
* Current treatment with topiramate, memantine, or barbiturates within two weeks of randomization
* Daytime use of benzodiazepines
* Current treatment with monoamine oxidase inhibitors within 4 weeks of randomization
* Treatment with a vagal nerve stimulator, ECT or deep brain stimulation within two weeks of randomization
* Psychosis other than psychotic experiences congruent with depressed mood during a period of depression
* Insulin-dependent diabetes or non-insulin dependent diabetes that is poorly controlled
* Other major medical disorder unless cleared by a study physician
* History of violence unless cleared by Dr. Driesen or Dr. Krystal because of extenuating circumstances. For example, an individual whose violent behavior was always coupled with substance abuse and had obtained stable sobriety with no violent incidents or an individual who had received successful pharmacotherapy for impulse control difficulties may be included.
* Individual meets criteria for a diagnosis of substance or alcohol use disorder within the three months prior to screening date. Individuals who meet criteria for mild alcohol use disorder within three months prior to screening date may be included in the study at investigator discretion. The diagnosis of mild alcohol use disorder shall be per DSM-5 and involve 2-3 symptoms. The PI's discretion will be based on the symptoms that are reported. The purpose of including individuals with mild alcohol use disorder is to extend recruitment to more individuals who can participate safely in the trial.
* A positive on screening urine drug test or, at the study physicians' discretion, on any drug screens given before the scans.
* A positive screening breathalyzer test or, at the study physicians' discretion, on any breathalyzer test given before the scans. This applies to all subjects, including those who make criteria for current mild alcohol use disorder.
* A 12-lead ECG at screening has clinically significant abnormalities as determined by the physician reading the ECG.
* Abnormality on clinical chemistry or hematology examination at the pre-study medical screening. Subjects with laboratory parameters outside the reference range for this age group will only be included if the study physician considers that such findings will not introduce additional risk factors.
* History of positive HIV or Hepatitis B
* Has received either prescribed or over-the-counter (OTC) centrally active medicine or herbal supplements within the week prior to the MRI scan. Subjects who have taken OTC medication or herbal supplements may still be entered into the study, if, in the opinions of the Principal/Co-Investigator, the medication received will not interfere with the study procedures or compromise safety.
* Known sensitivity to ketamine or heparin
* Resting blood pressure lower than 85/55 or higher than 140/90, or resting heart rate lower than 45/min or higher than 100/min, unless cleared by study physician. If a subject meets these blood pressure entrance criteria, but is being treated for high blood pressure, the study team will check with the subject's primary care physician or treatment provider to confirm that the subject is stable and normotensive on their current treatment plan.
* History of general intellectual disability
* History of claustrophobia
* Any clinically significant impairment of color vision or visual acuity after correction available in the scanner
* Presence of cardiac pacemaker or other electronic device or ferromagnetic metal foreign bodies in vulnerable positions as assessed by a Yale Magnetic Resonance Research Center standard pre-MRI screening questionnaire
* Subjects will be advised not to drive or operate heavy machinery for at least 24 hours after completing the infusion.
* Donation of blood in excess of 500 mL within 56 days prior to dosing or similar loss of blood due to other causes.
* Potential participants may be eliminated at the discretion of Dr. Krystal, Dr. Driesen, or the study physician.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Prefrontal functional connectivity | During ketamine infusion, approximately 2.5 hours
  This outcome will be assessed via functional magnetic resonance imaging (fMRI).
Cerebral metabolic rate of oxygen (CMRO2) | During ketamine infusion, approximately 2.5 hours.
  This outcome will be assessed via fMRI.

SECONDARY OUTCOMES:
Clinical improvement. | 24 hours post-infusion
  This outcome will be assessed by the Hamilton Depression Inventory, a clinician-rated instrument.

CONTACTS AND LOCATIONS:
Overall Officials: John Krystal, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No